CLINICAL TRIAL: NCT07030686
Title: Association Between Exercise, Patient-Reported Outcomes, and Clinical Events in Adult Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-101
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Survivorship; Recurrent; Recurrence; Cancer; Remission
Keywords: Survivorship; Exercise; cancer survivor; adult cancer survivor; no evidence of disease; 20-101; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Recurrence; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Usual Care
- Arm 2: Exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise following completion of active treatment for the primary index cancer
  Groups: Arm 2: Exercise

SUMMARY:
This protocol is a retrospective study using observational data to conduct a target trial emulation to examine the association of exercise on cancer specific endpoints and other clinical outcomes in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

Target trial (ideal RCT)

* Adult (≥18 years of age) patients with history of primary invasive cancer under surveillance at Memorial Sloan Kettering Cancer Center (MSK).
* Completion of an exercise survey (baseline) as part of MSK Cancer Survivorship Program and completion of a historical survey in the MSK Cancer Survivorship Program 9-15 months (time th) prior reporting non-exercising status [i.e., reporting <10 metabolic equivalent-hours per week (MET-h/week)]. Patients completing an additional exercise survey between th and baseline are excluded.
* No evidence of recurrent or metastatic disease in the 15 months prior to the baseline exercise assessment
* Completion of all definitive primary adjuvant therapy (e.g., chemotherapy, radiotherapy, targeted therapy) at least 3 months prior to completion of the historical exercise survey in a MSK Cancer Survivorship Program. Adjuvant hormonal therapy is permitted at any time.
* Undergoing surveillance in the Cancer Survivorship Program at MSK

Emulation using observational data

* Adult (≥18 years of age) cancer survivors under surveillance at Memorial Sloan Kettering Cancer Center (MSK) between 2011 and 2023.
* Assessment of self-reported exercise status via completion of an exercise survey as part of MSK Cancer Survivorship Program standard intake (baseline assessment).
* Non-exercising (i.e., reporting <5 MET-h/week) via completion of an exercise survey as part of MSK Cancer Survivorship Program standard intake 9-15 months prior to the baseline exercise assessment (historical exercise survey).
* Documented history of the following absolute contraindications to moderate-intensity exercise at any time prior to the baseline exercise assessment, assessed using the Elixhauser ICD codes: Congestive heart failure, valvular disease, chronic pulmonary disease, or renal failure.
* No evidence of recurrent or metastatic disease via radiological or pathological in EMR in the 15 months prior to the baseline exercise assessment.
* Completion of all definitive primary adjuvant therapy (e.g., chemotherapy, radiotherapy, targeted therapy) at least 3 months prior to completion of historical exercise survey (i.e., at least 3 months prior to t-1) as part of MSK Cancer Survivorship Program standard intake. Adjuvant endocrine therapy is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years of age) cancer survivors under surveillance at Memorial Sloan Kettering Cancer Center (MSK) between 2011 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Distant disease-free survival (DDFS) | 5 years
  To estimate the association of exercise vs. usual care (control) with Distant disease-free survival (DDFS) among patients following the completion of active treatment for the primary index cancer being monitored at MSK.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - City of Hope Cancer Center (Data Analysis Only), Duarte, California
  - University of California, Los Angeles (Data or Specimen Analysis Only), Los Angeles, California
  - Weill Cornell Medical College (Data or Specimen Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org